CLINICAL TRIAL: NCT01199510
Title: Efficacy Evaluation of SYSTANE® ULTRA in Patients Scheduled for Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMA-09-05
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye; Cataract Surgery
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care plus FID 112903 (Experimental): SYSTANE® ULTRA Lubricant Eye Drops dosed 4 times daily
  Interventions: Other: FID 112903 (SYSTANE® ULTRA Lubricant Eye Drops) plus standard of care
- Standard of Care only (Active Comparator): Post Cataract Standard of Care Regimen
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: FID 112903 (SYSTANE® ULTRA Lubricant Eye Drops) plus standard of care — Patients will dose 4 times daily for 30 days with FID 112903 and follow routine standard of care post-operatively
  Arms: Standard of Care plus FID 112903
Other: Standard of Care — Post Cataract Surgery Standard of Care
  Arms: Standard of Care only

SUMMARY:
The purpose of this study is to evaluate the effectiveness of FID 112903 (SYSTANE ULTRA® Lubricating Drops) plus standard of care to standard of care alone, in subjects with a history of intermittent eye irritation or dryness related to environmental factors and scheduled for routine cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age
* Patients must be seeking routine cataract extraction with monofocal intraocular lens implantation

Exclusion Criteria:

* Patients for whom both eyes do not meet all inclusion criteria and either eye meets any exclusion criteria.
* Patients cannot have a history of hypersensitivity to any component of FID 112903.
* Patients cannot have previous intraocular or corneal surgery or any planned within 30 days.
* Patients cannot use any ocular medications other than test article and standard of care post-op medications in past 14 days or during study.
* Patients cannot be on chronic systemic corticosteroid or other immunosuppressive therapy.
* Patients cannot have a history of steroid-responsive rise in intraocular pressure, glaucoma, or preoperative Intraocular pressure >25 millimeters mercury in either eye.
* Patients cannot have a history and/or current evidence of the following: clinically significant corneal scarring, blepharitis or macular pathology in either eye, Herpes zoster or Herpes simplex keratitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Ocular Comfort | 30 days
  Ocular comfort will be reported by the patient on a questionnaire

REFERENCES:
- [Result] http://www.escrs.org/abstracts/details.asp?confid=9&sessid=372&type=free&paperid=14295